CLINICAL TRIAL: NCT02529865
Title: Open-label, Multi-center, Single Arm Study to Evaluate the Efficacy and Safety of Periurethral Injection of Autologous Adipose Derived Regenerative Cells (ADRCs) for the Treatment of Male Stress Urinary Incontinence
Brief Title: Clinical Trial of Autologous Adipose Derived Regenerative Cells for the Treatment of Male Stress Urinary Incontinence
Acronym: ADRESU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, Momokazu Gotoh, MD, PhD, Professor at Department of Urology, Nagoya University Hospital, Nagoya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMCR-005; UMIN000017901 (Other: UMIN Clinical Trials Registry)
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Urinary Incontinence , Stress
Keywords: Cell Transplantation
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (1):
- ADRCs and Adipose tissue (Experimental): Periurethral injection of autologous adipose derived regenerative cells and adipose tissue
  Interventions: Biological: Periurethral injection of autologous ADRCs and adipose tissue

INTERVENTIONS:
Biological: Periurethral injection of autologous ADRCs and adipose tissue — 1 mL of the isolated ADRC is injected into the region of the external urethral sphincter, and another 4 mL of the ADRC and 16mL autologous adipose cells is injected under the urethral mucosa.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of periurethral injection of autologous Adipose Derived Regenerative Cells (ADRCs) in male stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Males with stress urinary incontinence with insufficient effect by behavioral therapy or pharmacotherapy persisting more than 1 year after either of the following surgical procedure:

  * Patients with symptoms after radical prostatectomy for localized prostate cancer and currently without relapse/metastasis, and PSA level less than 0.1 ng/mL for over 1 year
  * Patients with symptoms after transurethral prostatectomy or laser prostatectomy for prostatic hyperplasia, and PSA level less than 4.0 ng/mL over 1 year
* Age of 20 or above
* Mild to moderate urinary incontinence on the 24-hour pad test
* Patients who can keep a bladder diary in a satisfactory manner
* Patients who are willing and able to give signed consent

Exclusion Criteria:

* - Concurrent with any other types of urinary incontinence
* History of urinary or reproductive surgery within 6 months
* History of behavioral therapy or pharmacotherapy within 3 months
* Concurrent with diabetes insipidus
* History of radiotherapy in the lower urinary tract
* History of ADRCs treatment for stress urinary incontinence
* History of any type of cell therapy within 6 months
* Participation in any other clinical trial within 3 months
* Concurrent with lower urinary tract obstruction
* Concurrent with urolithiasis, urinary tract infection or interstitial cystitis
* History of recurrent urinary tract infection
* History of malignant neoplasm within 5 years or a suspicion of it
* Life expectancy of less than 1 year
* Any other patients whom the trial investigator deemed ineligible to this study

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients with improvement in urine leakage volume as greater than 50% reduction from baseline by 24-hour pad test | Baseline and 52 weeks (LOCF) after intervention

SECONDARY OUTCOMES:
Rate of patients with improvement in urine leakage volume as greater than 50% reduction from baseline by 24-hour pad test | Baseline, 2, 4, 12, 26, 38 and 52 weeks after intervention
Urine leakage volume by 24-hour pad test | Baseline, 2, 4, 12, 26, 38 and 52 weeks after intervention
Rate of patients with improvement in the number of incontinence episodes per day as greater than 50% reduction from baseline | Baseline, 2, 4, 12, 26, 38 and 52 weeks after intervention
Number of incontinence episodes per day | Baseline, 2, 4, 12, 26, 38 and 52 weeks after intervention
Number of pads used per day | Baseline, 2, 4, 12, 26, 38 and 52 weeks after intervention
QOL score (ICIQ-SF and KHQ) | Baseline, 26 and 52 weeks after intervention
Patient overall satisfaction | Baseline, 26 and 52 weeks after intervention
Urodynamic parameters (MUCP, FPL and ALPP) | Baseline, 2, 4, 12, 26 and 52 weeks after intervention
Blood flow at the injection site measured by transrectal ultrasonography | Baseline,12, 26 and 52 weeks after intervention
Injection site evaluated by pelvis MRI scan | Baseline, 2, 26 and 52 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Momokazu Gotoh, M.D., Ph.D., Principal Investigator — Department of Urology
Locations (4):
- Japan (4):
  - Nagoya university Hospital, Nagoya, Aichi-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Shinshu University Hospital, Matsumoto, Nagano
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi

REFERENCES:
- [Background] Shaw CF 3rd, Isab AA, Coffer MT, Mirabelli CK. Gold(I) efflux from auranofin-treated red blood cells. Evidence for a glutathione-gold-albumin metabolite. Biochem Pharmacol. 1990 Sep 15;40(6):1227-34. doi: 10.1016/0006-2952(90)90387-z. PMID 2403377
- [Background] Hersh WR, Greenes RA. Information retrieval in medicine: state of the art. MD Comput. 1990 Sep-Oct;7(5):302-11. PMID 2243546
- [Derived] Shimizu S, Yamamoto T, Nakayama S, Hirakawa A, Kuwatsuka Y, Funahashi Y, Matsukawa Y, Takanari K, Toriyama K, Kamei Y, Narimoto K, Yamanishi T, Ishizuka O, Mizuno M, Gotoh M. Design of a single-arm clinical trial of regenerative therapy by periurethral injection of adipose-derived regenerative cells for male stress urinary incontinence in Japan: the ADRESU study protocol. BMC Urol. 2017 Sep 25;17(1):89. doi: 10.1186/s12894-017-0282-7. PMID 28946874